CLINICAL TRIAL: NCT03779295
Title: Laser Therapy for Perioral Dermatitis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No subjects enrolled.
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Erica Ghareeb, Assistant Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1803028429
Record Dates: First submitted 2018-12-12; First posted 2018-12-19 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Perioral Dermatitis
Keywords: perioral dermatitis; laser therapy
MeSH Terms: conditions — Dermatitis, Perioral | interventions — Clindamycin

STUDY DESIGN:
Intervention Model Description: This will be a split face prospective trial. The face will be treated in halves. The halves will be randomized to receive topical clindamycin or PDL therapy and clindamycin. Both halves of the face will be treated with topical clindamycin. Per randomization, half of the face will be treated with pulse dye laser therapy at 595 nm, using 6.5 J/cm2, 10 mm spot size and a 6 millisecond pulse width.
Who Masked: Participant
Masking Description: The investigators will not remind the participant or other investigators which side of the face received laser therapy, however the investigators cannot completely "blind" either the participant or other investigators as they will be awake or performing the therapy, respectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Pulse laser therapy (Experimental): Pulse laser therapy will be randomly applied to right side or left side of face in addition to Clindamycin
  Interventions: Device: Pulse laser dye therapy (Device name: Candela Family of Pulsed Dye Laser Systems. 501k Number: K050673.); Drug: Clindamycin
- Clindamycin (Experimental): Clindamycin only applied to side of face that does not receive pulse laser therapy.
  Interventions: Drug: Clindamycin

INTERVENTIONS:
Device: Pulse laser dye therapy (Device name: Candela Family of Pulsed Dye Laser Systems. 501k Number: K050673.) — The face will be split and randomized, one half will receive pulsed laser dye therapy.
  Arms: Pulse laser therapy
Drug: Clindamycin — The entire face (both halves) will receive clindamycin.

SUMMARY:
Perioral dermatitis is an inflammation of the skin around the mouth. The cause of perioral dermatitis is unknown. Current treatment methods include oral antibiotics and topical calcenurin inhibitors, both of which produce side effects and have been relatively ineffective in the treatment of perioral dermatitis. The investigators hope to assess the efficacy of laser therapy in treatment of perioral dermatitis by using laser therapy on one half of the patients face and having patients apply topical medication (clindamycin) to their face for 8 weeks. The side of their face that receives laser therapy will be randomized. The investigators will assess the efficacy of laser therapy by counting the number of lesions that patients have before and after laser therapy, comparing photos of patient's perioral dermatitis before and after treatment, and having patient's rate their satisfaction of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* perioral dermatitis for greater than 1 month
* willing to return for follow-up visits 2 weeks, 4 weeks and 8 weeks following treatment.

Exclusion Criteria:

* skin type V or VI (due to risk of hyperpigmentation)
* pregnant
* breastfeeding
* unable to understand English
* mentally impaired
* incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
Change in number of lesions on side of the subject's face receiving laser therapy | initial study visit
  counting number of lesions on each side of the face
Change in number of lesions on side of the subject's face receiving laser therapy | 4 weeks
  counting number of lesions on each side of the face
Change in number of lesions on side of the subject's face receiving laser therapy | 8 weeks
  counting number of lesions on each side of the face
Change in number of lesions on side of the subject's face receiving clindamycin alone (NO laser therapy) | initial study visit
  counting number of lesions on each side of the face
Change in number of lesions on side of the subject's face receiving clindamycin alone (NO laser therapy) | 4 weeks
  counting number of lesions on each side of the face
Change in number of lesions on side of the subject's face receiving clindamycin alone (NO laser therapy) | 8 weeks
  counting number of lesions on each side of the face

SECONDARY OUTCOMES:
Patient opinion of side that improved more | 4 weeks
  Patients will grade satisfaction of treatment by answering "Which side of their face improved more from treatment?" with the option of responding "the right side/the left side/they are the same."
Patient opinion of side that improved more | 8 weeks
  Patients will grade satisfaction of treatment by answering "Which side of their face improved more from treatment?" with the option of responding "the right side/the left side/they are the same."

CONTACTS AND LOCATIONS:
Locations (1):
- West Virginia University University Town Centre Dermatology Clinic, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No